CLINICAL TRIAL: NCT01409018
Title: Pharmacokinetics of Itraconazole in Pediatric Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Oncology team, Janssen Korea Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH-R-0804
Record Dates: First submitted 2011-07-08; First posted 2011-08-03 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Pediatric, Cancer
Keywords: pediatric; cancer; invasive fungal disease; antifungal agent
MeSH Terms: conditions — Neoplasms; Invasive Fungal Infections | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Itraconazole (Experimental)
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — pharmacokinetics
  Other Names: Itraconazole(spranox)

SUMMARY:
This study investigated repeated-dose pharmacokinetics and safety of itraconazole and its active metabolite hydroxyitraconazole in pediatric cancer patients at risk for the development of invasive fungal disease.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who are under chemotherapy, and receive itraconazole.

Exclusion Criteria:

1. Patients with significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases.

   * Heart : fractional shortening < 30%, ejection fraction < 45%
   * Liver : total bilirubin ≥ 2 x upper limit of normal (ULN) ; aminotransferase ≥ 3 x ULN
   * Kidney : creatinine ≥ 2 x normal or GFR ≤ 60㎖/min/1.73㎡
2. Patients with hypersensitivity to azoles.
3. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
4. Pregnant or nursing women.
5. Psychiatric disorder that would preclude compliance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To investigate repeated-dose pharmacokinetics of itraconazole and its active metabolite hydroxyl itraconazole in pediatric cancer patients | 28 days
  1. Itraconazole administration 1) Oral for prophylaxis: 2mg/kg/dose,q12hr 2) IV for empirical therapy : After more than 2 days of oral prophylaxis, patients with persistent neutropenic fever / Induction : 5 mg/kg/dose, q12hr X 4 doses / Maintenance : 5 mg/kg/dose,q24hr
  2. Sampling 1) During oral : prior to the 5th dose 2) During IV : prior to the every induction and 1-5th maintenance doses, and 1, 2, 4, 8, 12, 24hr after the 3rd IV maintenance
  3. Analysis of drug concentrations : Plasma concentrations of itraconazole and hydroxyl-itraconazole are measured using HPLC.

SECONDARY OUTCOMES:
To assess empirical antifungal efficacy and safety in pediatric cancer patients | 28 days
  1. Efficacy evaluation : Treatment is considered successful if all five of the following criteria are met : treatment of baseline fungal infection, absence of breakthrough fungal infection, survival for 7 days after completion, resolution of fever (<38°C for 48hrs) in neutropenia, and no premature discontinuation because of drug related toxicity or lack of efficacy.
  2. Safety evaluation : Laboratory are performed at the time of enrollment, twice weekly during therapy, and 1 week after the end of therapy. Drug-related toxicity was graded according to the NCI Common Toxicity Criteria (v4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, M.D, ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea